CLINICAL TRIAL: NCT03663582
Title: A 24-Week Safety, Efficacy, Pharmacokinetic Study of Teduglutide in Japanese Subjects With Short Bowel Syndrome Who Are Dependent on Parenteral Support
Brief Title: Study of Teduglutide in Japanese Participants With Short Bowel Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHP633-306
Record Dates: First submitted 2018-08-28; First posted 2018-09-10 (Actual); Results first posted 2020-08-04 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome | interventions — teduglutide; Syringes; Needles

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Teduglutide 0.05 mg (Experimental): Participants will receive teduglutide 0.05 milligram per kilogram (mg/kg) subcutaneous (SC) injection once daily into 1 of the 4 quadrants of the abdomen or either thigh or arm for 24 weeks.
  Interventions: Drug: Teduglutide; Device: Syringe; Device: Needle; Device: Vial Adapter for Device

INTERVENTIONS:
Drug: Teduglutide — Teduglutide 0.05 mg/kg SC injection will be administered once daily into 1 of the 4 quadrants of the abdomen or either thigh or arm.
Device: Syringe — Teduglutide will be administered using syringe. Syringe is approved for use in Japan by Pharmaceuticals and Medical Devices Agency (PMDA).
Device: Needle — Teduglutide will be administered using needle. Needle is approved for use in Japan by PMDA.
Device: Vial Adapter for Device — Vial adapter for device is approved for use in Japan by PMDA.

SUMMARY:
The objectives of this clinical study are to evaluate the safety, efficacy, and pharmacokinetics (PK) of teduglutide in Japanese participants with short bowel syndrome (SBS) who are dependent on parenteral nutrition/intravenous (PN/IV) over a 24-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to voluntarily provide written, signed, and informed consent to participate in the study.
2. Male or female 16 years of age or older at the time of signing informed consent.
3. Intestinal failure due to short bowel syndrome (SBS) as a result of major intestinal resection (example, due to injury, volvulus, vascular disease, cancer, Crohn's disease) that resulted in at least 12 continuous months of parenteral nutrition/intravenous (PN/IV) dependence at the time of informed consent.
4. Parenteral nutrition requirement of at least 3 times per week during the week before the screening visit and during the 2 weeks prior to the baseline visit.
5. Stable PN/IV requirement for at least 4 consecutive weeks immediately prior to the start of teduglutide treatment. Stability is defined as: a. Actual PN/IV usage is similar to prescribed PN/IV; b. Baseline (Visit 2) 48-hour oral fluid intake and urine output (I/O) volumes fall within +/- 25 percent (%) of the respective 48-hour I/O volumes at the last optimization visit; c. Urine output volume should NOT fall below 2 liter (L) and should not exceed 4 L per 48 hours at the last optimization visit, the stabilization visit, and the baseline visit.
6. For participants with a history of Crohn's disease, clinical remission for at least 12 weeks prior to the baseline visit as demonstrated by clinical assessment, which may include procedure-based evidence of remission.
7. Females of childbearing potential must agree to comply with the contraceptive requirements of the protocol.
8. An understanding, ability, and willingness to fully comply with study procedures and restrictions.

Exclusion Criteria:

1. Participation in a clinical study using an experimental drug within 30 days or 5.5 halflives, whichever is longer, prior to screening, or concurrent participation in any other clinical study.
2. Use of glucagon-like peptide (GLP)-2 or human growth hormone or analogs of these hormones within the past 6 months.
3. Use of octreotide, GLP-1 analogs, dipeptidyl peptidase-IV inhibitors, or enteral glutamine within 30 days.
4. Previous use of teduglutide.
5. Participants with active inflammatory bowel disease (IBD) or participants with IBD who received a change in immunosuppressant therapy (example, azathioprine, anti- tumor necrosis factor (TNFs)) within the past 6 months.
6. Intestinal malabsorption due to a genetic condition, such as cystic fibrosis, microvillus inclusion disease, familial adenomatous polyposis, etc.
7. Chronic intestinal pseudo-obstruction or severe dysmotility.
8. Clinically significant intestinal stenosis or obstruction, or evidence of such on upper gastrointestinal (GI) series with small bowel follow-through, within the past 6 months.
9. Major GI surgical intervention, including bowel lengthening procedures, within the past 3 months (insertion of feeding tube or endoscopic procedure is allowed).
10. Unstable cardiac disease, (example, congestive heart failure, cyanotic disease, or congenital heart disease).
11. Moderate or severe renal impairment, defined as creatinine clearance less than (<) 50 millilitre (ml)/ minute (min).
12. Currently diagnosed with cancer or a history of any cancer except surgically curative skin cancer within the past 5 years.
13. Severe hepatobiliary disease including: a. Total bilirubin level greater than or equal to (>=) 2 times the upper limit of normal (ULN); b. Aspartate aminotransferase (AST) >=5 times ULN; c. Alanine aminotransferase (ALT) >=5 times ULN.
14. Active clinically significant pancreatic disease, including clinical signs of pancreatitis associated with elevations in serum amylase or lipase >=2 times ULN.
15. More than 4 SBS-related or PN/IV-related hospital admissions (example, central line associated bloodstream infection, bowel obstruction, severe fluid/electrolyte disturbances) within the past 12 months.
16. Unscheduled hospitalization within 30 days prior to screening.
17. Pregnant or lactating female.
18. Any condition or circumstance that in the investigator's opinion put the participant at any undue risk, prevent completion of the study, or interfere with analysis of the study results.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-07-06 (Actual); Primary Completion 2019-08-06 (Actual); Study Completion 2019-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (5):
- Japan (5):
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Hyogo College of Medicine Hospital, Hyōgo
  - Tohoku University Hospital, Miyagi-Ken
  - Osaka University Hospital, Osaka
  - Yokohama Municipal Citizen's Hospital, Yokohama

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be re-identified (due to the limited number of study participants/study sites, …).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 5 sites in Japan between 06 July 2018 (first participant first visit) and 06 August 2019 (last participant last visit).
Pre-assignment Details: A total of 7 participants were enrolled and received the treatment. Out of them, 6 participants completed the study.
Groups:
- Teduglutide: Participants received 0.05 milligram per kilogram (mg/kg) of teduglutide subcutaneous (SC) injection once daily into 1 of the 4 quadrants of the abdomen or either thigh or arm for 24 weeks.
Period: Overall Study
Arm/Group | Teduglutide
Started | 7
Completed | 6
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants in the intent-to-treat (ITT) population who received at least 1 dose of study treatment.
Arm/Group | Teduglutide
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.4 (8.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Weekly Parenteral Support (PS) Volume at End of Treatment/Early Termination (EOT/ET)
Description: Change from baseline in weekly PS volume at EOT/ET was reported.
Time Frame: Baseline, EOT/ET (up to Week 28)
Population: ITT population included all participants who were deemed eligible for teduglutide treatment at the baseline visit.
Measure: Mean (Standard Deviation); unit: Liter per week (L/Week)
Arm/Group | Teduglutide
Number analyzed (Participants) | 7
Liter per week (L/Week) | -2.92 (3.463)

2. Primary Outcome: Percent Change From Baseline in Weekly Parenteral Support (PS) Volume at End of Treatment/Early Termination (EOT/ET)
Description: Percent change from baseline in weekly PS volume at EOT/ET was reported.
Time Frame: Baseline, EOT/ET (up to Week 28)
Population: ITT population included all participants who were deemed eligible for teduglutide treatment at the baseline visit.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Teduglutide
Number analyzed (Participants) | 7
Percent change | -22.19 (24.953)

3. Primary Outcome: Percentage of Participants Who Achieved at Least 20 Percent (%) Reduction From Baseline in Weekly Parenteral Support (PS) Volume at Week 20
Description: Percentage of participants who achieved at least 20% reduction from baseline in weekly PS volume at Week 20 was reported.
Time Frame: Baseline, Week 20
Population: ITT population included all participants who were deemed eligible for teduglutide treatment at the baseline visit. Here, number of participants analyzed refer to the number of participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Teduglutide
Number analyzed (Participants) | 6
Percentage of participants | 66.7

4. Primary Outcome: Percentage of Participants Who Achieved at Least 20 Percent (%) Reduction From Baseline in Weekly Parenteral Support (PS) Volume at Week 24
Description: Percentage of participants who achieved at least 20% reduction from baseline in weekly PS volume at Week 24 was reported.
Time Frame: Baseline, Week 24
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Teduglutide
Number analyzed (Participants) | 6
Percentage of participants | 66.7

5. Primary Outcome: Percentage of Participants Who Achieved at Least 20 Percent (%) Reduction From Baseline in Weekly Parenteral Support (PS) at End of Treatment/Early Termination (EOT/ET)
Description: Percentage of participants who achieve at least 20% reduction from baseline in weekly PS at EOT/ET was reported.
Time Frame: Baseline, EOT/ET (up to Week 28)
Population: ITT population included all participants who were deemed eligible for teduglutide treatment at the baseline visit.
Measure: Number; unit: Percentage of participants
Arm/Group | Teduglutide
Number analyzed (Participants) | 7
Percentage of participants | 57.1

6. Primary Outcome: Change From Baseline in Days Per Week of Parenteral Support (PS) at End of Treatment/Early Termination (EOT/ET)
Description: Change from baseline in days per week of PS at EOT/ET was reported.
Time Frame: Baseline, EOT/ET (up to Week 28)
Population: ITT population included all participants who were deemed eligible for teduglutide treatment at the baseline visit.
Measure: Mean (Standard Deviation); unit: Days per Week
Arm/Group | Teduglutide
Number analyzed (Participants) | 7
Days per Week | -0.43 (1.134)

7. Primary Outcome: Change From Baseline in Plasma Citrulline Levels at End of Treatment/Early Termination (EOT/ET)
Description: Plasma citrulline levels were measured as a biomarker of enterocyte mass. Change from baseline in plasma citrulline levels up to EOT/ET was reported.
Time Frame: Baseline, EOT/ET (up to Week 28)
Population: ITT population included all participants who were deemed eligible for teduglutide treatment at the baseline visit.
Measure: Mean (Standard Deviation); unit: Micromoles (mcmol)
Arm/Group | Teduglutide
Number analyzed (Participants) | 7
Micromoles (mcmol) | 11.973 (11.7309)

8. Primary Outcome: Number of Participants Who Were Completely Weaned Off Parenteral Support (PS) at Week 24/End of Treatment (EOT)
Description: Number of participants who were completely weaned off PS at Week 24/EOT was reported.
Time Frame: Week 24/EOT
Population: ITT population included all participants who were deemed eligible for teduglutide treatment at the baseline visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Teduglutide
Number analyzed (Participants) | 7
Participants
  Weaned Off Parenteral Support: No | 7
  Weaned Off Parenteral Support: Yes | 0

9. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Zero to the Last Measurable Concentration (AUC0-t) of Teduglutide
Description: AUC0-t of teduglutide was reported.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10 and 12 hours Post-dose on Day 1; Pre-dose, 1, 2 hours Post-dose on Week 4 or Week 12
Population: Pharmacokinetic (PK) population included all participants who received at least 1 dose of teduglutide and had at least 1 evaluable post-dose pharmacokinetic concentration value.
Measure: Mean (Standard Deviation); unit: Hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Teduglutide
Number analyzed (Participants) | 7
Hour*nanogram per milliliter (h*ng/mL) | 240.3 (80.651)

10. Primary Outcome: Maximum Plasma Concentration (Cmax) of Teduglutide
Description: Cmax of teduglutide was reported.
Time Frame: as for outcome 9
Population: PK population included all participants who received at least 1 dose of teduglutide and had at least 1 evaluable post-dose pharmacokinetic concentration value.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Teduglutide
Number analyzed (Participants) | 7
Nanograms per milliliter (ng/mL) | 49.50 (16.427)

11. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) of Teduglutide
Description: Tmax of teduglutide was reported.
Time Frame: as for outcome 9
Population: as for outcome 10
Measure: Median (Full Range); unit: Hour
Arm/Group | Teduglutide
Number analyzed (Participants) | 7
Hour | 3.00 [1.87 to 5.92]

12. Primary Outcome: Terminal-phase Half-life (T1/2) of Teduglutide
Description: T1/2 of teduglutide was reported.
Time Frame: as for outcome 9
Population: PK population included all participants who received at least 1 dose of teduglutide and had at least 1 evaluable post-dose pharmacokinetic concentration value. Here, the number of participants analyzed refer to the number of participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: Hour
Arm/Group | Teduglutide
Number analyzed (Participants) | 6
Hour | 1.09 [0.751 to 1.30]

13. Primary Outcome: Apparent Clearance (CL/F) of Teduglutide
Description: CL/F of teduglutide was reported.
Time Frame: as for outcome 9
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Milliliter per hour (mL/h)
Arm/Group | Teduglutide
Number analyzed (Participants) | 6
Milliliter per hour (mL/h) | 10858.9 (4038.5)

14. Primary Outcome: Apparent Volume of Distribution (Vz/F) of Teduglutide
Description: Vz/F of teduglutide was reported.
Time Frame: as for outcome 9
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Milliliter (mL)
Arm/Group | Teduglutide
Number analyzed (Participants) | 6
Milliliter (mL) | 17167.4 (8371.9)

15. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. TEAEs were defined as AEs whose onset occurred, severity worsened, or intensity increased after receiving the study medication.
Time Frame: From start of study drug administration up to EOT/ET (up to Week 28)
Population: Safety population included all participants in the ITT population who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Teduglutide
Number analyzed (Participants) | 7
Participants | 7

16. Primary Outcome: Number of Participants With Clinically Significant Abnormalities in 12-Lead Electrocardiogram (ECG)
Description: 12-lead ECG was performed at the study center after the participant has been resting for at least 5 minutes. Number of participants with clinically significant abnormalities in 12-Lead ECG was reported.
Time Frame: From start of study drug administration up to EOT/ET (up to Week 28)
Population: Safety population included all participants in the ITT population who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Teduglutide
Number analyzed (Participants) | 7
Participants | 0

17. Primary Outcome: Change From Baseline in Blood Pressure at End of Treatment/Early Termination (EOT/ET)
Description: Change from baseline in systolic and diastolic blood pressure at EOT/ET was reported.
Time Frame: Baseline, EOT/ET (up to Week 28)
Population: Safety population included all participants in the ITT population who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Millimetre of mercury (mmHg)
Arm/Group | Teduglutide
Number analyzed (Participants) | 7
Millimetre of mercury (mmHg)
  Systolic Blood Pressure: EOT (up to Week 28) | 2.4 (19.37)
  Diastolic Blood Pressure: EOT (up to Week 28) | 6.6 (20.59)

18. Primary Outcome: Change From Baseline in Pulse Rate at End of Treatment/Early Termination (EOT/ET)
Description: Change from baseline in pulse rate at EOT/ET was reported.
Time Frame: Baseline, EOT/ET (up to Week 28)
Population: Safety population included all participants in the ITT population who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Beats per minute (beats/min)
Arm/Group | Teduglutide
Number analyzed (Participants) | 7
Beats per minute (beats/min) | 2.6 (9.88)

19. Primary Outcome: Change From Baseline in Body Temperature at End of Treatment/Early Termination (EOT/ET)
Description: Change from baseline in body temperature at EOT/ET was reported.
Time Frame: Baseline, EOT/ET (up to Week 28)
Population: Safety population included all participants in the ITT population who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Teduglutide
Number analyzed (Participants) | 7
Degree Celsius | -0.03 (0.411)

20. Primary Outcome: Change From Baseline in Hemoglobin at End of Treatment/Early Termination (EOT/ET)
Description: Change from baseline in hemoglobin at EOT/ET was reported.
Time Frame: Baseline, EOT/ET (up to Week 28)
Population: Safety population included all participants in the ITT population who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Gram per liter (g/L)
Arm/Group | Teduglutide
Number analyzed (Participants) | 7
Gram per liter (g/L) | -3.9 (12.94)

21. Primary Outcome: Change From Baseline in Hematocrit at End of Treatment/Early Termination (EOT/ET)
Description: Change from baseline in hematocrit at EOT/ET was reported.
Time Frame: Baseline, EOT/ET (up to Week 28)
Population: Safety population included all participants in the ITT population who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Volume per volume (v/v)
Arm/Group | Teduglutide
Number analyzed (Participants) | 7
Volume per volume (v/v) | -0.014 (0.0355)

22. Primary Outcome: Change From Baseline in Serum Blood Urea Nitrogen (BUN) at End of Treatment/Early Termination (EOT/ET)
Description: Change from baseline in serum blood urea nitrogen at EOT/ET was reported.
Time Frame: Baseline, EOT/ET (up to Week 28)
Population: Safety population included all participants in the ITT population who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Teduglutide
Number analyzed (Participants) | 7
mmol/L | 0 (0)

23. Primary Outcome: Change From Baseline in Creatinine at End of Treatment/Early Termination (EOT/ET)
Description: Change from baseline in creatinine at EOT/ET was reported.
Time Frame: Baseline, EOT/ET (up to Week 28)
Population: Safety population included all participants in the ITT population who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Micromoles per liter (mcmol/L)
Arm/Group | Teduglutide
Number analyzed (Participants) | 7
Micromoles per liter (mcmol/L) | -5.6 (8.42)

24. Primary Outcome: Change From Baseline in Urine Sodium at End of Treatment/Early Termination (EOT/ET)
Description: Change from baseline in urine sodium at EOT/ET was reported.
Time Frame: Baseline, EOT/ET (up to Week 28)
Population: Safety population included all participants in the ITT population who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Teduglutide
Number analyzed (Participants) | 7
millimoles per liter (mmol/L) | -2.1 (64.92)

25. Primary Outcome: Number of Participants Who Reported Positive Specific Antibodies to Teduglutide at End of Treatment/Early Termination (EOT/ET)
Description: Number of participants who reported positive specific antibodies to teduglutide at EOT/ET was reported.
Time Frame: EOT/ET (up to Week 28)
Population: Safety population included all participants in the ITT population who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Teduglutide
Number analyzed (Participants) | 7
Participants | 1

26. Primary Outcome: Change From Baseline in 48-Hour Urine Output at End of Treatment/Early Termination (EOT/ET)
Description: Change from baseline in 48-hour urine output at EOT/ET was reported.
Time Frame: Baseline, EOT/ET (up to Week 28)
Population: Safety population included all participants in the ITT population who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Milliliter per day (mL/day)
Arm/Group | Teduglutide
Number analyzed (Participants) | 7
Milliliter per day (mL/day) | 213.57 (242.757)

27. Primary Outcome: Change From Baseline in Body Weight at End of Treatment/Early Termination (EOT/ET)
Description: Change from baseline in body weight at EOT/ET was reported.
Time Frame: Baseline, EOT/ET (up to Week 28)
Population: Safety population included all participants in the ITT population who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | Teduglutide
Number analyzed (Participants) | 7
kilogram (kg) | 0.164 (1.1146)

28. Primary Outcome: Change From Baseline in Body Mass Index (BMI) at End of Treatment/Early Termination (EOT/ET)
Description: Change from baseline in BMI at EOT/ET was reported.
Time Frame: Baseline, EOT/ET (up to Week 28)
Population: Safety population included all participants in the ITT population who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Kilograms per square meter (kg/m^2)
Arm/Group | Teduglutide
Number analyzed (Participants) | 7
Kilograms per square meter (kg/m^2) | 0.07 (0.441)

29. Primary Outcome: Number of Participants With Abnormal Clinically Significant Changes in Gastrointestinal (GI) Specific Tests at Week 24/ET (Early Termination)
Description: GI specific tests included colonoscopy or sigmoidoscopy, abdominal ultrasound, upper GI series with small bowel follow-through (UGI/SBFT). Number of participants with abnormal clinically significant changes in gastrointestinal specific tests at Week 24/ET was reported.
Time Frame: Week 24/ET
Population: Safety population included all participants in the ITT population who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Teduglutide
Number analyzed (Participants) | 7
Participants | 0

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to EOT/ET (up to Week 28)
Arm/Group | Teduglutide
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 3/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teduglutide (N=7)
Device related infection (Infections and infestations) | 1 (1)
Medical device site infection (Infections and infestations) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teduglutide (N=7)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Polycythaemia (Blood and lymphatic system disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Injection site reaction (General disorders) | 2 (2)
Pyrexia (General disorders) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 (1)
Muscle contusion (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Hypozincaemia (Metabolism and nutrition disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2018-09-27): https://cdn.clinicaltrials.gov/large-docs/82/NCT03663582/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-13): https://cdn.clinicaltrials.gov/large-docs/82/NCT03663582/SAP_001.pdf